CLINICAL TRIAL: NCT02796339
Title: A Phase-II Clinical Trial on the Effectiveness of a Nutritional Supplement With Natural Mastiha in Inflammatory Bowel Diseases Patients.
Brief Title: A Study on the Effectiveness of a Nutritional Supplement With Natural Mastiha in Inflammatory Bowel Diseases.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, "Assistant Professor in Foods & Human Nutrition", Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Mastiha IBD-GR (304)
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; natural Mastiha; supplement
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — mastiha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mastiha (Active Comparator): This arm of patients will receive natural Mastiha supplements at the dosage of 2.8g daily. Patients with active disease will be administered with supplements for 3 months, whereas patients in remission will be administered with supplements for 6 months.
  Interventions: Dietary Supplement: Mastiha
- Placebo (Placebo Comparator): This arm of patients will receive placebo . Patients with active disease will be administered with placebo for 3 months, whereas patients in remission will be administered with placebo for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mastiha
  Arms: Mastiha
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of a supplement with natural Mastiha on Inflammatory Bowel Diseases (IBD). U.S. Food and Drug Administration has classified Mastiha as GRAS. Previous research demonstrates Mastiha's safety, as well as anti-inflammatory, antimicrobial and antioxidant properties. In addition, the European Medicine Agency has recently recognized Mastiha as a natural medicine and classified it to the category of traditional herbal medicines in diarrhea problems, mild dyspeptic disorders, skin inflammation and healing (EMA/HMPC/46758/2015). Since IBD is a chronic disease characterized by inflammation and oxidative stress and based on previous small-scale studies, the present study aims at demonstrating the effectiveness of this supplement adjunct to the conservative treatment of IBD.

To this end, confirmed IBD patients, with distinguished Ulcerative Colitis (UC) and Crohn's Disease (CD) will be enrolled based on certain inclusion and exclusion criteria. The staff of the study will provide detailed information regarding the aims, the methods, anticipated benefits and potential hazards of the study and all patients will receive the Patient Information Leaflet (PIL). Ample time (48 hours) will be provided in order to decide whether they want to participate in the protocol. Each patient agreeing to participate will sign an Informed Consent document and the staff will explain to patients that they are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason. A copy of the signed Informed Consent will be given to the participant.

100 IBD patients will be allocated to either Mastiha or placebo group. The Mastiha group will receive natural Mastiha supplement at a dose of 2.8 g daily while placebo group will receive respectively placebo. The intervention will last 3 months for patients in relapse and 6 months for patients in remission. They will receive all the supplements they will consume during the intervention at the start of the trial. Both groups will continue their medical treatment, which must be unaltered throughout the trial. Additionally, all patients will receive standard nutritional advice by dieticians and will be encouraged to report any adverse effects they may experience during the intervention. The trial will be blinded in all implicated persons; neither the staff of the trial nor the patients will be aware of which kind intervention they receive.

Patients are assessed after randomisation according to the following tools:

* Medical history
* Dietary history
* Harvey & Bradshaw Activity Index Assessment
* Mayo Activity Index assessment
* Anthropometric data measurement: body weight (kg), height (cm), Body Mass Index (kg/m2)
* Inflammatory Bowel Disease Questionnaire
* DNA isolation from whole blood.
* Biochemical measurements: Complete blood count, albumin, lipid profile, glucose, electrolytes, liver enzymes, amylase, fibrinogen.
* Evaluation of inflammation in serum samples. Circulating serum levels of IL-6, IL-8, IL-17A, IL-17F, IL-18, IL-21, IL-22, TL1A, TGF-β, ICAM-1, MADCAM-1 and E-selectin are measured), in all active CD and UC patients. Inflammatory markers are also estimated in stool samples: calprotectin, lactoferrin and lysozyme,
* Oxidative stress assessment in serum/plasma samples. Oxidised LDL, serum oxidisability and F2-isoprostanes are quantified.
* Detection of metabolites and complete metabolomic profile in plasma samples.
* Stool samples collection for the assessment of gut microbiota in active patients.
* Genetic and epigenetic profile

Subsequent assessments: There is a biweekly telephone contact with the patients to monitor compliance and side effects. At the end of the intervention each subject undergoes the baseline assessment.

ELIGIBILITY:
Eligibility criteria for patients in relapse

Inclusion criteria:

* Age 18-67 years
* Active disease, CD defined by Harvey & Bradshaw Activity Index ≥4; UC defined by Partial Mayo Clinic Score (2<= Mayo Scoring Index)
* Childbearing age with a negative pregnancy test at eligibility and baseline assessment
* Stable treatment with steroids for at least 2 weeks before the start of the trial, mesalamine and mesalamine analogues for 4 weeks and immunosuppressants for 8 weeks
* Stable medication during the whole period of the 3-month intervention

Exclusion criteria:

* Positive stool culture for enteric pathogens or Clostridium difficile toxin
* Antibiotic treatment during and 2 months prior to screening
* Bowel surgery ≤3 months prior to screening; a planned elective surgery or hospitalisation during the study; clinically significant short bowel syndrome; presence of an intra-abdominal abscess or a fistula with clinical or radiological evidence of an associated abscess; ileostomy; colostomy
* Enteral or parenteral nutrition; Alcohol or drug abuse,Vitamin or inorganic supplements, vegan or macrobiotic diet before and during the trial
* Any malignancy in the year prior to screening; CVD; peptic ulcer
* Pregnancy, lactation

Eligibility criteria for patients in remission

Inclusion criteria:

* Age 18-67 years
* Inactive disease (>3 months), CD defined by Harvey & Bradshaw (<6 Index) and UC defined by Partial Mayo Clinic (0-1 Mayo Scoring Index)
* Biochemical remission
* Childbearing age with a negative pregnancy test at eligibility and baseline assessment
* Stable treatment with azathioprine or mesalamine and mesalamine analogues
* Stable medication during the whole period of the 6-month intervention

Exclusion criteria:

* Positive stool culture for enteric pathogens or Clostridium difficile toxin
* Antibiotic treatment during and 2 months prior to screening
* Bowel surgery ≤3 months prior to screening; a planned elective surgery or hospitalisation during the study; clinically significant short bowel syndrome; presence of an intra-abdominal abscess or a fistula with clinical or radiological evidence of an associated abscess; ileostomy; colostomy
* Enteral or parenteral nutrition; Alcohol or drug abuse
* Vitamin or inorganic supplements, vegan or macrobiotic diet before and during the trial
* Any malignancy in the year prior to screening; CVD; peptic ulcer
* Pregnancy, lactation

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | Change in IBDQ will be assessed at 3 months from baseline in active IBD patients and at 6 months in inactive IBD patients. Data will be presented through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Objective symptoms questionnaire (rectal bleeding and stool frequency, visible blood in faeces and urgency). | Change in objective symptoms will be assessed at 3 months from baseline in active IBD patients and at 6 months in inactive IBD patients. Data will be presented through study completion, an average of 1 year.
C-reactive protein (CRP) | Change in CRP will be assessed at 3 months from baseline in active IBD patients and at 6 months in inactive IBD patients. Data will be presented through study completion, an average of 1 year.
Lab inflammatory biomarkers through sandwich Elisa assays. | Change in lab inflammatory biomarkers will be assessed at 3 months from baseline in active IBD patients and at 6 months in inactive IBD patients. Data will be presented through study completion, an average of 1 year.
Subjective symptoms questionnaire (physician rating of disease activity) | Change in subjective symptoms will be assessed at 3 months from baseline in active IBD patients and at 6 months in inactive IBD patients. Data will be presented through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: ANDRIANA KALIORA, AS.PROFESSOR, Principal Investigator — ASS.PROFESSOR
Locations (1):
- Harokopio University, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksoy A, Duran N, Koksal F. In vitro and in vivo antimicrobial effects of mastic chewing gum against Streptococcus mutans and mutans streptococci. Arch Oral Biol. 2006 Jun;51(6):476-81. doi: 10.1016/j.archoralbio.2005.11.003. Epub 2005 Dec 15. PMID 16343417
- [Background] Al-Habbal MJ, Al-Habbal Z, Huwez FU. A double-blind controlled clinical trial of mastic and placebo in the treatment of duodenal ulcer. Clin Exp Pharmacol Physiol. 1984 Sep-Oct;11(5):541-4. doi: 10.1111/j.1440-1681.1984.tb00864.x. PMID 6395994
- [Background] Al-Said MS, Ageel AM, Parmar NS, Tariq M. Evaluation of mastic, a crude drug obtained from Pistacia lentiscus for gastric and duodenal anti-ulcer activity. J Ethnopharmacol. 1986 Mar;15(3):271-8. doi: 10.1016/0378-8741(86)90165-0. PMID 3724207
- [Background] Appleyard CB, Hernandez G, Rios-Bedoya CF. Basic epidemiology of inflammatory bowel disease in Puerto Rico. Inflamm Bowel Dis. 2004 Mar;10(2):106-11. doi: 10.1097/00054725-200403000-00007. PMID 15168809
- [Background] Assimopoulou AN, Papageorgiou VP. GC-MS analysis of penta- and tetra-cyclic triterpenes from resins of Pistacia species. Part I. Pistacia lentiscus var. Chia. Biomed Chromatogr. 2005 May;19(4):285-311. doi: 10.1002/bmc.454. PMID 15651084
- [Background] Assimopoulou AN, Papageorgiou VP. GC-MS analysis of penta- and tetra-cyclic triterpenes from resins of Pistacia species. Part II. Pistacia terebinthus var. Chia. Biomed Chromatogr. 2005 Oct;19(8):586-605. doi: 10.1002/bmc.484. PMID 15770609
- [Background] Bjerrum JT, Wang Y, Hao F, Coskun M, Ludwig C, Gunther U, Nielsen OH. Metabonomics of human fecal extracts characterize ulcerative colitis, Crohn's disease and healthy individuals. Metabolomics. 2015;11:122-133. doi: 10.1007/s11306-014-0677-3. Epub 2014 Jun 1. PMID 25598765
- [Background] Bountziouka V, Bathrellou E, Giotopoulou A, Katsagoni C, Bonou M, Vallianou N, Barbetseas J, Avgerinos PC, Panagiotakos DB. Development, repeatability and validity regarding energy and macronutrient intake of a semi-quantitative food frequency questionnaire: methodological considerations. Nutr Metab Cardiovasc Dis. 2012 Aug;22(8):659-67. doi: 10.1016/j.numecd.2010.10.015. Epub 2011 Jan 26. PMID 21269818
- [Background] Burisch J, Munkholm P. Inflammatory bowel disease epidemiology. Curr Opin Gastroenterol. 2013 Jul;29(4):357-62. doi: 10.1097/MOG.0b013e32836229fb. PMID 23695429
- [Background] Chang S, Malter L, Hudesman D. Disease monitoring in inflammatory bowel disease. World J Gastroenterol. 2015 Oct 28;21(40):11246-59. doi: 10.3748/wjg.v21.i40.11246. PMID 26523100
- [Background] Chapman CG, Pekow J. The emerging role of miRNAs in inflammatory bowel disease: a review. Therap Adv Gastroenterol. 2015 Jan;8(1):4-22. doi: 10.1177/1756283X14547360. PMID 25553076
- [Background] Cleynen I, Boucher G, Jostins L, Schumm LP, Zeissig S, Ahmad T, Andersen V, Andrews JM, Annese V, Brand S, Brant SR, Cho JH, Daly MJ, Dubinsky M, Duerr RH, Ferguson LR, Franke A, Gearry RB, Goyette P, Hakonarson H, Halfvarson J, Hov JR, Huang H, Kennedy NA, Kupcinskas L, Lawrance IC, Lee JC, Satsangi J, Schreiber S, Theatre E, van der Meulen-de Jong AE, Weersma RK, Wilson DC; International Inflammatory Bowel Disease Genetics Consortium; Parkes M, Vermeire S, Rioux JD, Mansfield J, Silverberg MS, Radford-Smith G, McGovern DP, Barrett JC, Lees CW. Inherited determinants of Crohn's disease and ulcerative colitis phenotypes: a genetic association study. Lancet. 2016 Jan 9;387(10014):156-67. doi: 10.1016/S0140-6736(15)00465-1. Epub 2015 Oct 18. PMID 26490195
- [Background] Cohen LB, Nanau RM, Delzor F, Neuman MG. Biologic therapies in inflammatory bowel disease. Transl Res. 2014 Jun;163(6):533-56. doi: 10.1016/j.trsl.2014.01.002. Epub 2014 Jan 7. PMID 24467968
- [Background] de Cassia da Silveira e Sa R, Andrade LN, de Sousa DP. A review on anti-inflammatory activity of monoterpenes. Molecules. 2013 Jan 18;18(1):1227-54. doi: 10.3390/molecules18011227. PMID 23334570
- [Background] Duda-Chodak A, Tarko T, Satora P, Sroka P. Interaction of dietary compounds, especially polyphenols, with the intestinal microbiota: a review. Eur J Nutr. 2015 Apr;54(3):325-41. doi: 10.1007/s00394-015-0852-y. Epub 2015 Feb 12. PMID 25672526
- [Background] Franchimont D, Vermeire S, El Housni H, Pierik M, Van Steen K, Gustot T, Quertinmont E, Abramowicz M, Van Gossum A, Deviere J, Rutgeerts P. Deficient host-bacteria interactions in inflammatory bowel disease? The toll-like receptor (TLR)-4 Asp299gly polymorphism is associated with Crohn's disease and ulcerative colitis. Gut. 2004 Jul;53(7):987-92. doi: 10.1136/gut.2003.030205. PMID 15194649
- [Background] Georgiadis I, Karatzas T, Korou LM, Agrogiannis G, Vlachos IS, Pantopoulou A, Tzanetakou IP, Katsilambros N, Perrea DN. Evaluation of Chios mastic gum on lipid and glucose metabolism in diabetic mice. J Med Food. 2014 Mar;17(3):393-9. doi: 10.1089/jmf.2013.0069. Epub 2014 Jan 9. PMID 24404977
- [Background] Giaginis C, Theocharis S. Current evidence on the anticancer potential of Chios mastic gum. Nutr Cancer. 2011 Nov;63(8):1174-84. doi: 10.1080/01635581.2011.607546. Epub 2011 Nov 1. PMID 22044444
- [Background] Gioxari A, Kaliora AC, Papalois A, Agrogiannis G, Triantafillidis JK, Andrikopoulos NK. Pistacia lentiscus resin regulates intestinal damage and inflammation in trinitrobenzene sulfonic acid-induced colitis. J Med Food. 2011 Nov;14(11):1403-11. doi: 10.1089/jmf.2010.0240. Epub 2011 May 25. PMID 21612460
- [Background] Gonzalez-Burgos E, Gomez-Serranillos MP. Terpene compounds in nature: a review of their potential antioxidant activity. Curr Med Chem. 2012;19(31):5319-41. doi: 10.2174/092986712803833335. PMID 22963623
- [Background] Huwez FU, Al-Habbal MJ. Mastic in treatment of benign gastric ulcers. Gastroenterol Jpn. 1986 Jun;21(3):273-4. doi: 10.1007/BF02774571. No abstract available. PMID 3732760
- [Background] Kaliora AC, Stathopoulou MG, Triantafillidis JK, Dedoussis GV, Andrikopoulos NK. Alterations in the function of circulating mononuclear cells derived from patients with Crohn's disease treated with mastic. World J Gastroenterol. 2007 Dec 7;13(45):6031-6. doi: 10.3748/wjg.v13.45.6031. PMID 18023095
- [Background] Kaliora AC, Stathopoulou MG, Triantafillidis JK, Dedoussis GV, Andrikopoulos NK. Chios mastic treatment of patients with active Crohn's disease. World J Gastroenterol. 2007 Feb 7;13(5):748-53. doi: 10.3748/wjg.v13.i5.748. PMID 17278198
- [Background] Kottakis F, Kouzi-Koliakou K, Pendas S, Kountouras J, Choli-Papadopoulou T. Effects of mastic gum Pistacia lentiscus var. Chia on innate cellular immune effectors. Eur J Gastroenterol Hepatol. 2009 Feb;21(2):143-9. doi: 10.1097/MEG.0b013e32831c50c9. PMID 19212203
- [Background] Koutsoudaki C, Krsek M, Rodger A. Chemical composition and antibacterial activity of the essential oil and the gum of Pistacia lentiscus Var. chia. J Agric Food Chem. 2005 Oct 5;53(20):7681-5. doi: 10.1021/jf050639s. PMID 16190616
- [Background] Loddo I, Romano C. Inflammatory Bowel Disease: Genetics, Epigenetics, and Pathogenesis. Front Immunol. 2015 Nov 2;6:551. doi: 10.3389/fimmu.2015.00551. eCollection 2015. PMID 26579126
- [Background] Morgan XC, Tickle TL, Sokol H, Gevers D, Devaney KL, Ward DV, Reyes JA, Shah SA, LeLeiko N, Snapper SB, Bousvaros A, Korzenik J, Sands BE, Xavier RJ, Huttenhower C. Dysfunction of the intestinal microbiome in inflammatory bowel disease and treatment. Genome Biol. 2012 Apr 16;13(9):R79. doi: 10.1186/gb-2012-13-9-r79. PMID 23013615
- [Background] Papalois A, Gioxari A, Kaliora AC, Lymperopoulou A, Agrogiannis G, Papada E, Andrikopoulos NK. Chios mastic fractions in experimental colitis: implication of the nuclear factor kappaB pathway in cultured HT29 cells. J Med Food. 2012 Nov;15(11):974-83. doi: 10.1089/jmf.2012.0018. Epub 2012 Aug 14. PMID 22891614
- [Background] Paraschos S, Magiatis P, Mitakou S, Petraki K, Kalliaropoulos A, Maragkoudakis P, Mentis A, Sgouras D, Skaltsounis AL. In vitro and in vivo activities of Chios mastic gum extracts and constituents against Helicobacter pylori. Antimicrob Agents Chemother. 2007 Feb;51(2):551-9. doi: 10.1128/AAC.00642-06. Epub 2006 Nov 20. PMID 17116667
- [Background] Sakagami H, Kishino K, Kobayashi M, Hashimoto K, Iida S, Shimetani A, Nakamura Y, Takahashi K, Ikarashi T, Fukamachi H, Satoh K, Nakashima H, Shimizu T, Takeda K, Watanabe S, Nakamura W. Selective antibacterial and apoptosis-modulating activities of mastic. In Vivo. 2009 Mar-Apr;23(2):215-23. PMID 19414406
- [Background] Sands BE. Biomarkers of Inflammation in Inflammatory Bowel Disease. Gastroenterology. 2015 Oct;149(5):1275-1285.e2. doi: 10.1053/j.gastro.2015.07.003. Epub 2015 Jul 9. PMID 26166315
- [Background] Triantafyllou A, Bikineyeva A, Dikalova A, Nazarewicz R, Lerakis S, Dikalov S. Anti-inflammatory activity of Chios mastic gum is associated with inhibition of TNF-alpha induced oxidative stress. Nutr J. 2011 Jun 6;10:64. doi: 10.1186/1475-2891-10-64. PMID 21645369